CLINICAL TRIAL: NCT02165137
Title: Quality Control in the Management of Major Trauma Patients at Aarau Cantonal Hospital - Evaluation of Processes and Patient Outcome
Brief Title: Management of Major Trauma Patients at Aarau Trauma Center - Evaluation of Processes and Patient Outcome
Status: Completed | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Collaborators: Kantonsspital Aarau, Wissenschaftlicher Fond (Unknown); Suva (Unknown)
Responsible Party: Principal Investigator, Thomas Gross, MD, Prof. Dr. med., Kantonsspital Aarau
Other Study IDs: 2012-008; 2012-008 (Other: Kantonale Ethikkommission AG/ SO)
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Injury; Trauma; Major Trauma; Multiple Trauma
Keywords: trauma; major trauma; multiple trauma; outcome; quality; process Management; emergency room; trauma center
MeSH Terms: conditions — Wounds and Injuries; Multiple Trauma; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- trauma patients: type and severity of patients, circumstances and trauma pre- and post-injury / -quality initiative

SUMMARY:
Quality control and improvement project: Assessment and analysis of processes and outcome in trauma emergency room and major trauma patients at the Aarau trauma center (cantonal hospital) with regard to initial emergency management, hospital processes and short- and long-term (1-and 2-year) outcome of patients (subjective and objective). Comparison of processes and outcome pre- and post- project initiative. Benchmarking with the literature and by participation in the German and Swiss Trauma registry each.

DETAILED DESCRIPTION:
Registry of all emergency patients arriving at Aarau trauma center following trauma with regard to possibly injury related pre- and inhospital demographic factors, process variables and outcome Parameters.

ELIGIBILITY:
Inclusion Criteria:

* major trauma: New Injury Severity Score (NISS) >=8
* for longer-term outcome: only patients firm in German language and able to respond to the postal questionnaire by themselves

Exclusion Criteria:

* no Trauma
* injury >24h before arrival at Aarau Cantonal Hospital
* NISS<8
* for longer-term outcome: patients not firm in German language and not able to respond to the postal questionnaire by themselves (dead, unavailable, refusal to participate, dementia, age<16 years ecc.); a categorising compilation of cases is supposed to exclude any possible study bias

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All emergency patients treated at Aarau Cantonal Hospital following trauma (<24h postinjury) with suspected major trama
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Actual)
Dates: Start 2010-01; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
emergency room process times | hours (<6)

SECONDARY OUTCOMES:
hospital mortality | 30 days
Euro Quality of Life Group health-related quality of life on five dimensions (EQ-5D) | 1 and 2 year follow-up
  score
Trauma Outcome Profile (TOP) | 1 and 2 year follow-up
  score
Quality of Life after Brain Injury (QOLIBRI) | 1 and 2 year follow-up
  score
medical outcomes study Short Form-36 (SF-36) | 1 and 2 year follow-up
  score
reduced capacity to work | 1 and 2 year outcome
  Value (%);e.g. see Gross T, Attenberger C, Huegli RW, Amsler F. Factors associated with reduced longer-term capacity to work in patients after polytrauma: a Swiss trauma center experience. J Am Coll Surg. 2010 Jul;211(1):81-91

OTHER OUTCOMES:
invalidity | at least 4 year post-injury
  % of disability to work (i.e., basis for resulting amount of insurance pension)
insurance payments | at least 4 years post-injury
  Swiss Francs

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gross, MD, Prof., Principal Investigator — Aarau Cantonal Hospital
Locations (1):
- Aarau Cantonal Hospital, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Gross T, Amsler F. Prevalence and incidence of longer term pain in survivors of polytrauma. Surgery. 2011 Nov;150(5):985-95. doi: 10.1016/j.surg.2011.04.003. Epub 2011 Jun 15. PMID 21676423
- [Background] Attenberger C, Amsler F, Gross T. Clinical evaluation of the Trauma Outcome Profile (TOP) in the longer-term follow-up of polytrauma patients. Injury. 2012 Sep;43(9):1566-74. doi: 10.1016/j.injury.2011.01.002. Epub 2011 Jan 20. PMID 21255778
- [Background] Gross T, Attenberger C, Huegli RW, Amsler F. Factors associated with reduced longer-term capacity to work in patients after polytrauma: a Swiss trauma center experience. J Am Coll Surg. 2010 Jul;211(1):81-91. doi: 10.1016/j.jamcollsurg.2010.02.042. Epub 2010 May 15. PMID 20610253
- [Background] Fueglistaler P, Amsler F, Schuepp M, Fueglistaler-Montali I, Attenberger C, Pargger H, Jacob AL, Gross T. Prognostic value of Sequential Organ Failure Assessment and Simplified Acute Physiology II Score compared with trauma scores in the outcome of multiple-trauma patients. Am J Surg. 2010 Aug;200(2):204-14. doi: 10.1016/j.amjsurg.2009.08.035. Epub 2010 Mar 15. PMID 20227058
- [Background] Fuglistaler-Montali I, Attenberger C, Fuglistaler P, Jacob AL, Amsler F, Gross T. In search of benchmarking for mortality following multiple trauma: a Swiss trauma center experience. World J Surg. 2009 Nov;33(11):2477-89. doi: 10.1007/s00268-009-0193-1. PMID 19693630
- [Background] Gross T, Schuepp M, Attenberger C, Pargger H, Amsler F. Outcome in polytraumatized patients with and without brain injury. Acta Anaesthesiol Scand. 2012 Oct;56(9):1163-74. doi: 10.1111/j.1399-6576.2012.02724.x. Epub 2012 Jun 26. PMID 22735047
- [Result] Gross T, Morell S, Scholz SM, Amsler F. The capacity of baseline patient, injury, treatment and outcome data to predict reduced capacity to work and accident insurer costs - a Swiss prospective 4-year longitudinal trauma centre evaluation. Swiss Med Wkly. 2019 Dec 17;149:w20144. doi: 10.4414/smw.2019.20144. eCollection 2019 Dec 16. PMID 31846504
- [Result] Gross T, Morell S, Amsler F. To What Extent Are Main Accident-Insurer Cases Representative of All Significantly Injured? A Swiss Monocenter Perspective. J Insur Med. 2019;48(1):65-78. doi: 10.17849/insm-48-1-1-14.1. Epub 2019 Apr 24. PMID 31017516
- [Result] Gross T, Morell S, Amsler F. Gender-Specific Improvements in Outcome 1 and 2 Years After Major Trauma. J Surg Res. 2019 Mar;235:459-469. doi: 10.1016/j.jss.2018.10.024. Epub 2018 Nov 21. PMID 30691830
- [Result] Gross T, Braken P, Amsler F. Trauma center need: the American College of Surgeons' definition in contrast to Swiss highly specialized medicine regulations-a Swiss trauma center perspective. Eur J Trauma Emerg Surg. 2020 Apr;46(2):397-406. doi: 10.1007/s00068-018-1027-3. Epub 2018 Oct 13. PMID 30317378
- [Result] Born K, Amsler F, Gross T. Prospective evaluation of the Quality of Life after Brain Injury (QOLIBRI) score: minor differences in patients with major versus no or mild traumatic brain injury at one-year follow up. Health Qual Life Outcomes. 2018 Jul 9;16(1):136. doi: 10.1186/s12955-018-0966-z. PMID 29986710
- [Result] Gross T, Amsler F. One-year outcome following brain injury: a comparison of younger versus elderly major trauma patients. Arch Orthop Trauma Surg. 2018 Oct;138(10):1375-1387. doi: 10.1007/s00402-018-2974-1. Epub 2018 Jun 11. PMID 29948226
- [Result] Gross T, Morell S, Amsler F. Longer-term quality of life following major trauma: age only significantly affects outcome after the age of 80 years. Clin Interv Aging. 2018 Apr 30;13:773-785. doi: 10.2147/CIA.S158344. eCollection 2018. PMID 29750022
- [Result] Braken P, Amsler F, Gross T. Simple modification of trauma mechanism alarm criteria published for the TraumaNetwork DGU(R) may significantly improve overtriage - a cross sectional study. Scand J Trauma Resusc Emerg Med. 2018 Apr 24;26(1):32. doi: 10.1186/s13049-018-0498-x. PMID 29690930
- [Result] Bundi M, Meier L, Amsler F, Gross T. [Impact of weather, time of day and season on the admission and outcome of major trauma patients]. Unfallchirurg. 2018 Jan;121(1):10-19. doi: 10.1007/s00113-016-0267-0. German. PMID 27778061
- [Result] Gross T, Amsler F. [Long-term outcome following multiple trauma in working age : A prospective study in a Swiss trauma center]. Unfallchirurg. 2016 Nov;119(11):921-928. doi: 10.1007/s00113-014-2720-2. German. PMID 25633852
- [Result] Gross T, Amsler F. [Emergency room and major trauma treatment is a "loss-making business" : A Swiss trauma center experience with current DRG reimbursement]. Unfallchirurg. 2021 Sep;124(9):747-754. doi: 10.1007/s00113-020-00937-w. Epub 2020 Dec 18. German. PMID 33337516
- [Result] Walkner S, Amsler F, Gross T. [How often is a chest tube needed following thoracic trauma in the severely injured-and when is more needed? : Data from a Swiss trauma center for planning of resources and surgical training]. Chirurg. 2021 Aug;92(8):721-728. doi: 10.1007/s00104-020-01292-7. German. PMID 33034700
- [Result] Gross T, Morell S, Amsler F. Medically graded reduced capacity to work (RCW) following significant injury as explained by patient related outcome measures (PROMs): A prospective trauma center evaluation. Disabil Health J. 2021 Oct;14(4):101114. doi: 10.1016/j.dhjo.2021.101114. Epub 2021 May 10. PMID 34059469
- [Result] Gross T, Amsler F. Main factors predicting somatic, psychological, and cognitive patient outcomes after significant injury: a pilot study of a simple prognostic tool. BJS Open. 2021 Nov 9;5(6):zrab109. doi: 10.1093/bjsopen/zrab109. PMID 34864883
- [Result] Zeindler M, Amsler F, Gross T. Comparative analysis of MGAP, GAP, and RISC2 as predictors of patient outcome and emergency interventional need in emergency room treatment of the injured. Eur J Trauma Emerg Surg. 2021 Dec;47(6):2017-2027. doi: 10.1007/s00068-020-01361-w. Epub 2020 Apr 13. PMID 32285143
- [Result] Fiumedinisi FA, Amsler F, Gross T. Short-term outcome following significant trauma: increasing age per se has only a relatively low impact. Eur J Trauma Emerg Surg. 2021 Dec;47(6):1979-1992. doi: 10.1007/s00068-020-01357-6. Epub 2020 Apr 16. PMID 32300851
- [Result] Magyar CTJ, Maeder F, Diepers M, Amsler F, Gross T. Detailed information gain and therapeutic impact of whole body computed tomography supplementary to conventional radiological diagnostics in blunt trauma emergency treatment: a consecutive trauma centre evaluation. Eur J Trauma Emerg Surg. 2022 Apr;48(2):921-931. doi: 10.1007/s00068-020-01502-1. Epub 2020 Sep 30. PMID 32997166